CLINICAL TRIAL: NCT06988020
Title: Evaluation of Optimised Whole-body MRI Examinations Incorporating "Pseudo-scanner" Sequences (ZTE, "Zero Echo Time" AND Lava Flex) for the Detection of Bone Lesions in Multiple Myeloma
Brief Title: "Pseudo-scanner" MRI Sequences for the Detection of Bone Lesions in Multiple Myeloma
Acronym: MM-ZTE-II
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: General Electric (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025/13FEV/071
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Multiple Myeloma Bone Disease
Keywords: bone; imaging; mri; multiple myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Whole body MRI (Other): There is only one cohort where each patient have the standard of care follow up (PET/CT) and Whole body MRI- ZTE sequence for the study
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — Whole body MRI including ZTE sequences

SUMMARY:
Recent work has confirmed the diagnostic performance of pseudo-CT sequences for detecting osteolytic lesions. Their integration into whole body MRI (WB MRI) could transform the diagnostic approach to MM, by allowing a combined assessment of bone marrow involvement, tissue viability and osteolysis, during a single non-irradiating imaging examination. Since the preliminary work mentioned above, optimizations have been made to the pseudo-CT sequences, including the addition of deep learning (correcting noise in the images) and the correction of chemical shift artifact (linked to the coexistence of hydrated tissue and fatty tissue), which carry real hope of improving their diagnostic potential and accuracy.

DETAILED DESCRIPTION:
Currently recommended imaging techniques for detecting bone lesions include whole-body MRI (WB-MRI), computed tomography (CT), and PET-CT. WB-MRI and PET-CT outperform CT for assessing treatment response, with WB-MRI already being the imaging modality of choice in many countries. However WB-MRI, the technique of choice for detecting bone marrow involvement, does not allow visualization of mineral bone, limiting its ability to accurately assess osteolysis. Zero Echo Time (ZTE) and Lava Flex Low Flip Angle (LF) MRI sequences represent a major advance, providing visualization of tissues at very short T2 relaxation times with resolution close to that of CT. These new sequences (known as pseudo-CT or pseudo-CT) offer for the first time the opportunity to study mineral bone by MRI, thus considerably increasing the diagnostic potential of this modality in MM.

ELIGIBILITY:
Inclusion Criteria:

Patient with newly diagnosed multiple myeloma, for whom bone imaging is required for staging.

* Recurrent patient after intensive treatment (high dose chemotherapy, bone marrow transplant, etc.).
* Patient requiring a PET / CT considered as the technique of choice in these stages of the disease.

Exclusion Criteria:

* Implanted material incompatible with MRI.
* Severe claustrophobia.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the diagnostic performance of the different imaging protocols | through study completion, an average of 1 year
  The diagnostic performance of the different imaging protocols will be evaluated by analyzing the receptor efficiency function (ROC curve) and by estimating the Sensitivity (Se), Specificity (Sp), Positive Predictive Value (PPV), Negative Predictive Value (NPV) ) as well as the Predictive Accuracy (Acc) of the different imaging protocols.

SECONDARY OUTCOMES:
Comparison of Sensitivity (Se) and Predictive Precision (Acc) of the different imaging protocols | through study completion, an average of 1 year
  McNemar test on paired data. The Gold Standard will be determined by a panel of independent experts based on all available imaging techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Lecouvet, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (2):
- Belgium (2):
  - Cliniques Universitaires Saint Luc, Brussels
  - Cliniques universitaires Saint-Luc, Brussels

IPD SHARING:
Plan to Share IPD: No
Ethic reason

REFERENCES:
- [Background] Lecouvet FE, Zan D, Lepot D, Chabot C, Vekemans MC, Duchene G, Chiabai O, Triqueneaux P, Kirchgesner T, Taihi L, Poujol J, Gheysens O, Michoux N. MRI-based Zero Echo Time and Black Bone Pseudo-CT Compared with Whole-Body CT to Detect Osteolytic Lesions in Multiple Myeloma. Radiology. 2024 Oct;313(1):e231817. doi: 10.1148/radiol.231817. PMID 39377681
- [Background] Lecouvet FE, Vande Berg BC, Malghem J, Maldague BE. Magnetic resonance and computed tomography imaging in multiple myeloma. Semin Musculoskelet Radiol. 2001;5(1):43-55. doi: 10.1055/s-2001-12920. PMID 11371335
- [Background] Lecouvet FE, Boyadzhiev D, Collette L, Berckmans M, Michoux N, Triqueneaux P, Pasoglou V, Jamar F, Vekemans MC. MRI versus 18F-FDG-PET/CT for detecting bone marrow involvement in multiple myeloma: diagnostic performance and clinical relevance. Eur Radiol. 2020 Apr;30(4):1927-1937. doi: 10.1007/s00330-019-06469-1. Epub 2019 Dec 16. PMID 31844960